CLINICAL TRIAL: NCT05070585
Title: Isothiocyanates and Metabolic Health
Acronym: IMH
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: The Swedish School of Sport and Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: SwedishSchoolSport
Record Dates: First submitted 2021-09-01; First posted 2021-10-07 (Actual); Last update posted 2022-12-06 (Actual); Status verified 2022-12

CONDITIONS: Metabolic Disturbance
Keywords: Isothiocyanates; Blood lactate; Glucose regulation; Nrf2

STUDY DESIGN:
Intervention Model Description: Randomized, placebo controlled, cross-over study
Who Masked: Participant, Investigator
Masking Description: The subjects will receive a sprout juice or a placebo juice made of alfalfa sprouts.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Isothiocyanate Rich Juice (Experimental): The juices will contain 37,5g isothiocyanate rich sprouts and be delivered frozen to the subjects. The subjects will be instructed to consume two juices per day.
  Interventions: Dietary Supplement: Isothiocyanate rich sprouts
- Placebo Juice (Placebo Comparator): The juices will contain 37,5g alfalfa sprouts and be delivered frozen to the subjects. The subjects will be instructed to consume two juices per day.
  Interventions: Dietary Supplement: Placebo Juice

INTERVENTIONS:
Dietary Supplement: Isothiocyanate rich sprouts — Isothiocyanate rich sprout juice consumption for 1 week
  Arms: Isothiocyanate Rich Juice
Dietary Supplement: Placebo Juice — Sprout juice devoid of isothiocyanates for 1 week
  Arms: Placebo Juice

SUMMARY:
Many sprouts, for example broccoli sprouts, contain substances that have shown to have protective effects, both against oxidative stress and against carcinogenic substances.

In this study we will investigate the activation of the body's antioxidant defense system and effect on blood lactate and glucose after 1 week of isothiocyanate rich sprout supplementation. The subjects will perform maximal and submaximal work test, blood sampling, muscle biopsies and blood pressure monitoring post supplementation. We hypothesize that 1 week of supplementation of isothiocyanate rich sprouts alters blood lactate and glucose metabolism and activates the body's antioxidant defense system.

DETAILED DESCRIPTION:
Many sprouts, for example broccoli sprouts, contain high levels of glucosinolates, which can be converted to the bioactive substances isothiocyanates. This conversion is assisted by another plant enzyme, myrosinase, which is released when the plant is mechanically processed. It is believed that this reaction is part of the plant's natural defense against pest insects and other animals that attack the plant in the early developmental stage. In cell and animal studies supplementation with isothiocyanates has been shown to induce the protein Nrf2 which is a so-called "Master regulator" of the body's antioxidant defenses and activates more than 200 genes that together provide a strong protection against oxidative and mutagenic stress.

In this study we will investigate Nrf2 activation in human skeletal muscle and effect on lactate-, glucose metabolism after 1 week of isothiocyanate rich sprout supplementation. The study is a double-blinded, randomized, placebo controlled, cross-over study with 4 weeks wash-out between the interventions. We will perform maximal- and submaximal work test and monitor blood glucose and lactate during the tests. Also, in the post intervention phases we will perform muscle biopsies, glucose tolerance tests and monitor blood pressure.

The hypothesis is that 1 week of isothiocyanate rich sprout supplementation activates Nrf2 in human skeletal muscle and alters blood lactate and glucose metabolism in rest and during exercise.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteer
* 18-45 years old

Exclusion Criteria:

* Any chronic disease
* Inability to perform cycling exercise
* Allergic to anesthesia

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2021-10-20 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2023-12-05 (Estimated)

PRIMARY OUTCOMES:
Blood lactate | Acute during sub maximal exercise
  Changes in blood lactate during exercise
Nrf2 activation | Acute after 1 week of supplementation
  Increased Nrf2 protein in human skeletal muscle
Glucose regulation | Throughout 1 week of supplementation
  Improved continuous glucose control

SECONDARY OUTCOMES:
Glucose tolerance test | 120 minutes
  Improved glucose regulation in rest
Clinic blood pressure | Acute after 1 week of supplementation
  Blood pressure regulation

CONTACTS AND LOCATIONS:
Locations (1):
- Swedish School of Sports and Health Sciences, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No